CLINICAL TRIAL: NCT04436601
Title: Effect of Polyethylene Glycol Versus Lactulose on Hepatic Encephalopathy in Patients With Liver Cirrhosis; a Randomized Clinical Trial (PEGHE Trial)
Brief Title: Polyethylene Glycol Versus Lactulose on Hepatic Encephalopathy in Patients With Cirrhosis;(PEGHE Trial)
Acronym: PEGHE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Om Parkash, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191002MED
Record Dates: First submitted 2020-05-23; First posted 2020-06-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Polyethylene Glycols; Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It would be a double blinded study. Investigator assessing the participants and following the patient will be masked to the allocation of treatment group. Participants would be masked to their treatment group as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactulose (Active Comparator): 90 ml of Lactulose dissolved in 750 ml of water administered orally by mouth or nasogastric tube (three doses within 24 hrs) continued up to 72 hours or until patient discharge, whichever comes first.
  Interventions: Drug: Lactulose
- PEG: Polyethylene Glycol (Experimental): Three or four sachet of Movicol(PEG) will be dissolved in 750 ml of water and will be given over 24 hrs as 3 doses orally by mouth or Nasogastric tube and will continue up to 72 hours or until patient discharge, whichever comes first
  Interventions: Drug: Polyethylene Glycols

INTERVENTIONS:
Drug: Polyethylene Glycols — Polyethylene glycol will be administered to half of the study patients, and their response recorded and compared with that of the Lactulose arm.
  Arms: PEG: Polyethylene Glycol
Drug: Lactulose — Lactulose (standard of care) will be administered to half of the study patients and their response recorded.
  Arms: Lactulose

SUMMARY:
Hepatic Encephaopathy is a common complication occurring in patients with Liver cirrhosis. Patients usually develop mild confusion, sleep disturbance or obtundation. It occurs due to accumulation of excess ammonia in the brain, as the liver is unable to metabolize the ammonia. The common gold standard treatment recommended for patients with Hepatic Encephalopathy is Lactulose syrup. This is a non absorbable sugar, often combined with an antibiotic called Rifaxamine to treat this condition.

Polyethylene glycol is in a class of medications called osmotic laxatives which works by causing water to be retained with the stool. PEG and lactulose, when used together, result in faster resolution of symptoms suggesting that PEG may be superior to standard lactulose therapy in these patients.

Non-absorbable sugars like lactulose are associated with non-serious (mainly gastrointestinal) adverse events like diarrhea and bloating Hence, due to the side effect profile, newer drugs continue to be tested for treatment of Hepatic Encephalopathy.

The aim of this research project is to compare the effect of PEG versus lactulose for treatment of HE in patients with liver cirrhosis. The investigators want to compare the resolution of HE as the main outcome. In addition, they will compare length of stay, non-serious (mainly gastrointestinal) adverse events, and 3 months outcome. The investigators hypothesize that rapid purgation of the gut using PEG may resolve HE more effectively than lactulose.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a common neuropsychiatric complication of liver cirrhosis manifested by mild confusion, sleep disturbance or obtundation. Lactulose treatment has long been the standard of care, which presumably acidifies stool and eradicates toxic metabolites. However a third of these patients with hepatic encephalopathy do not respond to this standard treatment and have refractory HE. Hence newer drugs with effective improvement in HE and better side effect profile are still being tested.

Polyethylene glycol (PEG) is in a class of medications called osmotic laxatives which works by causing water to be retained with the stool. PEG and lactulose, when used together, result in rapid overt HE resolution within 24 hours compared to the standard-of-care lactulose, suggesting that PEG may be superior to standard lactulose therapy in patients with cirrhosis hospitalized for acute HE.

Rationale Non-absorbable disaccharides like lactulose are associated with non-serious (mainly gastrointestinal) adverse events like diarrhea and bloating, hence, due to the side effect profile, newer drugs continue to be tested for treatment of HE.

Hypothesis and Aim The aim of this research project is to compare the effect of PEG with Lactulose for treatment of Hepatic Encephalopathy in patients with liver cirrhosis. The investigators want to compare the resolution of HE as the main outcome. In addition, they would compare length of stay, non-serious (mainly gastrointestinal) adverse events, and 3 months outcome. The investigators hypothesize that rapid purgation of the gut using PEG may resolve HE more effectively than lactulose.

These aims are original in that the investigators aim to test this hypothesis on a different patient population (South Asian), where the predominant cause of cirrhosis is due to viral hepatitis C and B. In addition,the investigators will also look at the effect of PEG v lactulose on 3 months outcome in this study.

Significance The significance of this proposal is that if the investigators can prove the hypothesis, it will add to the currently limited evidence on use of PEG in treatment of HE in the world. PEG might have a better side effect profile when compared to lactulose. Based on current market pricing of lactulose, if PEG is found to have favorable outcome then it might be more cost effective as well. Hence PEG might be a useful alternative in 30% of those who don't respond to lactulose, if PEG shows favorable outcome.

Objective Primary: To determine the effect of PEG versus Lactulose on resolution of HE in patients with liver cirrhosis during inpatient stay at 24 hours, 48 hours and 72 hours .

Secondary: To determine the effect of Lactulose versus PEG on length of stay, and 3 months outcome in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients of 18-80 years admitted to Aga Khan University Hospital
2. With Chronic liver disease: Chronic liver disease will be defined based on ultra-sonographic evidence of chronic liver disease including shrunken liver, dilated portal vein, splenomegaly.
3. With Hepatic encephalopathy; Hepatic encephalopathy will be defined as the onset of disorientation or asterixis according to The International Society for Hepatic Encephalopathy and Nitrogen Metabolism consensus and will be assessed using HESA score
4. Presence of first degree relative for consent (Next of kin)

Exclusion Criteria:

1. Allergy to PEG
2. Bowel obstruction or perforation diagnosed clinically or on Xray
3. Major psychiatric illness; on benzodiazepines
4. Treated with locally acting antibiotics (rifaximin) in the previous 7 days;
5. Active gastrointestinal tract bleeding
6. Acute Liver failure:defined as coagulopathy (international normalized ratio >1.5) with any degree of AMS in the absence of underlying chronic liver disease (CLD)
7. Female patients if pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of Hepatic Encephalopathy | Change in HESA score at 24 hours, 48 hours and if applicable, 72 hours of drug administration
  Calculated using Hepatic Encephalopathy scoring Algorithm (HESA). Resolution is defined as reduction of at least 1 grade of HESA score after 24 hours, 48 hours and if applicable 72 hours of therapy during hospital stay

SECONDARY OUTCOMES:
Mean Length of inpatient stay in hours | at time of patient discharge, an average of 72 hours
  Duration of hospital stay will be recorded in hours
3 months outcome (readmission with Hepatic Encephalopathy) | The three month outcome will be assessed at clinic follow-up at 3 month or by phone call if patient is lost to follow up
  Patient will be asked at 3 month follow up if there was any other readmission anywhere with Hepatic Encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Om Parkash, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Combined data, relevant to the study publication will be made available

REFERENCES:
- [Background] Poordad FF. Review article: the burden of hepatic encephalopathy. Aliment Pharmacol Ther. 2007 Feb;25 Suppl 1:3-9. doi: 10.1111/j.1746-6342.2006.03215.x. PMID 17295846
- [Background] Rahimi RS, Rockey DC. Novel Ammonia-Lowering Agents for Hepatic Encephalopathy. Clin Liver Dis. 2015 Aug;19(3):539-49. doi: 10.1016/j.cld.2015.04.008. Epub 2015 May 30. PMID 26195207
- [Background] Elkington SG, Floch MH, Conn HO. Lactulose in the treatment of chronic portal-systemic encephalopathy. A double-blind clinical trial. N Engl J Med. 1969 Aug 21;281(8):408-12. doi: 10.1056/NEJM196908212810803. No abstract available. PMID 4894464
- [Background] Sharma P, Sharma BC, Sarin SK. Predictors of nonresponse to lactulose in patients with cirrhosis and hepatic encephalopathy. Eur J Gastroenterol Hepatol. 2010 May;22(5):526-31. doi: 10.1097/MEG.0b013e3283341b7d. PMID 20009938
- [Background] Tapper EB, Jiang ZG, Patwardhan VR. Refining the ammonia hypothesis: a physiology-driven approach to the treatment of hepatic encephalopathy. Mayo Clin Proc. 2015 May;90(5):646-58. doi: 10.1016/j.mayocp.2015.03.003. Epub 2015 Apr 9. PMID 25865476
- [Background] Romero-Gomez M, Jover M, Del Campo JA, Royo JL, Hoyas E, Galan JJ, Montoliu C, Baccaro E, Guevara M, Cordoba J, Soriano G, Navarro JM, Martinez-Sierra C, Grande L, Galindo A, Mira E, Manes S, Ruiz A. Variations in the promoter region of the glutaminase gene and the development of hepatic encephalopathy in patients with cirrhosis: a cohort study. Ann Intern Med. 2010 Sep 7;153(5):281-8. doi: 10.7326/0003-4819-153-5-201009070-00002. PMID 20820037
- [Background] Jain L, Sharma BC, Sharma P, Srivastava S, Agrawal A, Sarin SK. Serum endotoxin and inflammatory mediators in patients with cirrhosis and hepatic encephalopathy. Dig Liver Dis. 2012 Dec;44(12):1027-31. doi: 10.1016/j.dld.2012.07.002. Epub 2012 Aug 9. PMID 22883217
- [Background] Wijdicks EF. Hepatic Encephalopathy. N Engl J Med. 2016 Oct 27;375(17):1660-1670. doi: 10.1056/NEJMra1600561. No abstract available. PMID 27783916
- [Background] Zuberi BF, Alvi H, Zuberi FF, Rasheed T, Nawaz Z, Fatima-Tuz-Zohra. Frequency of minimal hepatic encepalopathy in illeterate patients with compensated cirrhosis. Pak J Med Sci. 2016 May-Jun;32(3):595-8. doi: 10.12669/pjms.323.9655. PMID 27375696
- [Background] Gerber T, Schomerus H. Hepatic encephalopathy in liver cirrhosis: pathogenesis, diagnosis and management. Drugs. 2000 Dec;60(6):1353-70. doi: 10.2165/00003495-200060060-00008. PMID 11152016
- [Background] Gluud LL, Vilstrup H, Morgan MY. Non-absorbable disaccharides versus placebo/no intervention and lactulose versus lactitol for the prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2016 May 6;2016(5):CD003044. doi: 10.1002/14651858.CD003044.pub4. PMID 27153247
- [Background] Williams R, Bass N. Rifaximin, a nonabsorbed oral antibiotic, in the treatment of hepatic encephalopathy: antimicrobial activity, efficacy, and safety. Rev Gastroenterol Disord. 2005;5 Suppl 1:S10-8. PMID 15976747
- [Background] Kimer N, Krag A, Moller S, Bendtsen F, Gluud LL. Systematic review with meta-analysis: the effects of rifaximin in hepatic encephalopathy. Aliment Pharmacol Ther. 2014 Jul;40(2):123-32. doi: 10.1111/apt.12803. Epub 2014 May 21. PMID 24849268
- [Background] Rahimi RS, Singal AG, Cuthbert JA, Rockey DC. Lactulose vs polyethylene glycol 3350--electrolyte solution for treatment of overt hepatic encephalopathy: the HELP randomized clinical trial. JAMA Intern Med. 2014 Nov;174(11):1727-33. doi: 10.1001/jamainternmed.2014.4746. PMID 25243839
- [Background] Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Alexeeva O, Zupanets IA, Grinevich V, Baranovsky A, Dudar L, Fadieienko G, Kharchenko N, Klaryts'ka I, Morozov V, Grewal P, McCashland T, Reddy KG, Reddy KR, Syplyviy V, Bass NM, Dickinson K, Norris C, Coakley D, Mokhtarani M, Scharschmidt BF; HALT-HE Study Group. Randomized, double-blind, controlled study of glycerol phenylbutyrate in hepatic encephalopathy. Hepatology. 2014 Mar;59(3):1073-83. doi: 10.1002/hep.26611. PMID 23847109
- [Background] American Association for the Study of Liver Diseases; European Association for the Study of the Liver. Hepatic encephalopathy in chronic liver disease: 2014 practice guideline by the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases. J Hepatol. 2014 Sep;61(3):642-59. doi: 10.1016/j.jhep.2014.05.042. Epub 2014 Jul 8. No abstract available. PMID 25015420
- [Background] Gluud LL, Vilstrup H, Morgan MY. Non-absorbable disaccharides versus placebo/no intervention and lactulose versus lactitol for the prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2016 Apr 18;4:CD003044. doi: 10.1002/14651858.CD003044.pub3. PMID 27089005
- [Background] Shehata HH, Elfert AA, Abdin AA, Soliman SM, Elkhouly RA, Hawash NI, Soliman HH. Randomized controlled trial of polyethylene glycol versus lactulose for the treatment of overt hepatic encephalopathy. Eur J Gastroenterol Hepatol. 2018 Dec;30(12):1476-1481. doi: 10.1097/MEG.0000000000001267. PMID 30234645
- [Background] Naderian M, Akbari H, Saeedi M, Sohrabpour AA. Polyethylene Glycol and Lactulose versus Lactulose Alone in the Treatment of Hepatic Encephalopathy in Patients with Cirrhosis: A Non-Inferiority Randomized Controlled Trial. Middle East J Dig Dis. 2017 Jan;9(1):12-19. doi: 10.15171/mejdd.2016.46. PMID 28316761
- [Background] Friedman S, Schiano T. Cirrhosis and its sequelae. Cecil Textbook of Medicine 22nd ed Philadelphia, Pa: Saunders. 2004:936-44.
- [Background] American College of R. Expert Panel on Gastrointestinal Imaging. Liver lesion characterization Reston, Va: American College of Radiology. 2002.
- [Background] Hassanein TI, Hilsabeck RC, Perry W. Introduction to the Hepatic Encephalopathy Scoring Algorithm (HESA). Dig Dis Sci. 2008 Feb;53(2):529-38. doi: 10.1007/s10620-007-9895-0. Epub 2007 Aug 21. PMID 17710551
- [Background] Lee WM, Stravitz RT, Larson AM. Introduction to the revised American Association for the Study of Liver Diseases Position Paper on acute liver failure 2011. Hepatology. 2012 Mar;55(3):965-7. doi: 10.1002/hep.25551. No abstract available. PMID 22213561
- [Background] Mendez-Sanchez N, Aguilar-Ramirez JR, Reyes A, Dehesa M, Juorez A, Castneda B, Sanchez-Avila F, Poo JL, Guevara Gonzalez L, Lizardi J, Valdovinos MA, Uribe M, Contreras AM, Tirado P, Aguirre J, Rivera-Benitez C, Santiago-Santiago R, Bosques-Padilla F, Munoz L, Guerroro A, Ramos M, Rodriguez-Hernandez H, Jacobo-Karam J; Grupo de Estudio, Asociacion Mexicana de Hepatologia. Etiology of liver cirrhosis in Mexico. Ann Hepatol. 2004 Jan-Mar;3(1):30-3. PMID 15118577